CLINICAL TRIAL: NCT02355925
Title: Evaluation the Effect of Intrauterine Injection of Human Chorionic Gonadotropin Injection (hCG) Before Frozen Embryo Transfer on Implantation, Clinical Pregnancy and Miscarriage Rates: Double Blind Randomized Clinical Trial ,Phase 3
Brief Title: Intrauterine Injection of Human Chorionic Gonadotropin Injection (hCG) Before Frozen Embryo Transfer on Cycle Outcomes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: royan-Emb-020
Record Dates: First submitted 2015-01-27; First posted 2015-02-04 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2016-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- uhCG (Experimental): The patients who receive Intrauterine injection of 500 IU of uhCG (0.5ml) before embryo transfer
  Interventions: Drug: intrauterine injection of uhCG
- Placebo (Placebo Comparator): The patients who underwent Intrauterine injection of placebo (normal saline 0.5 ml) before embryo transfer
  Interventions: Drug: Placebo
- control (Other): the embryonic transfer is done without the intrauterine hCG injection. The ET procedure is performed just like in the other two groups.
  Interventions: Other: control

INTERVENTIONS:
Drug: intrauterine injection of uhCG — 40 μL of tissue culture medium (G.2plus ref. 10132, Vitrolife) containing either 500 IU of hCG (Choriomon®, IBSA SA, Switzerland) is injected intrauterine, approximately 7 minutes before embryo transfer.
  Arms: uhCG
Drug: Placebo — only 40 μL of tissue culture medium (G.2plus ref. 10132, Vitrolife) is injected intrauterine, approximately 7 minutes before embryo transfer.
  Arms: Placebo
Other: control — the embryonic transfer is done without the intrauterine hCG injection. The ET procedure is performed just like in the other two groups.
  Arms: control

SUMMARY:
The present study is designed as a pilot study with 150 patients in each group. Data collection form will be filled by the researcher who does not know the type of intervention in each group. Data analysis will be done through descriptive and perceptive statistical methods by using SPSS software version 20 for windows

DETAILED DESCRIPTION:
This randomized double blinded clinical trial is conducted to evaluate the effect of intrauterine injection of human chorionic gonadotropin (hCG) before frozen embryo transfer (ET). The study protocol is approved by the Ethics Committee (Institutional Review Board) of Royan institute. The study is performed according to the Declaration of Helsinki for medical research. All participants provide informed consent after explaining the purpose of the study. All the patients with primary infertility who have only one fresh implantation failure and undergoing frozen embryo transfer cycles are enrolled. In all patients, endometrial preparation is performed by hormonal replacement method. In this way, endometrial preparation is started from the second or third day of menstrual cycle with daily administration of 6 mg oral estradiol valerate (Estraval®, Aburaihan CO, Tehran, Iran) for 8 days. After 8 days of estradiol administration, if favourable thickness of endometrium (≥ 8 mm) is confirmed by ultrasound, estradiol valerate is continued with the same dose and 50 mg progesterone (Progestin®, Aburaihan Pharmaceutical. Co., Tehran, Iran) intramuscularly is administered for 3 days and then embryos are transferred. Otherwise the dosage of estradiol is increased to 8 mg/day until the favourable thickness of endometrium be achieved. In the Embryo transfer day, the eligible patients are randomized using sealed opaque envelopes into three groups. In all study groups, the patient is put in the lithotomy position, and the cervix is visualized using Cusco's speculum. The cervical mucous is wiped out using a sterile piece of gauze, and then the mucous is partially removed by gentle suction with a 1-mL syringe. Embryo transfer is performed using a soft catheter (Labotec, Gottingen Germany). After the catheter is passed the internal cervical os; in group A (experimental group) 40 μL of tissue culture medium (G.2plus ref. 10132, Vitrolife) containing either 500 IU of hCG (Choriomon®, IBSA SA, Switzerland) is injected intrauterine. In group B (the placebo group) only 40 μL of tissue culture medium (G.2plus ref. 10132, Vitrolife) is injected intrauterine. In both groups, approximately 7 minutes after injection, the embryos are loaded into another ET catheter and are transferred into the uterine cavity. In group C (the control group), the ET is done without the intrauterine hCG injection. The ET procedure is performed just like in the other two groups.

According to the patients' age, up to 3 frozen-thawed Embryos are thawed and transferred at cleavage stage. Hormone therapy is continued until pregnancy test (2 weeks after ET) is performed and in case of positive pregnancy, administration of estradiol valerate and progesterone continued by 10 and 12 weeks of gestation. Chemical pregnancy is defined by a rising hCG level in serum without the detection of a gestational sac. Clinical pregnancy is diagnosed by the presence of a gestational sac with fetal heart in vaginal ultrasonography. The miscarriage rate is defined as the loss of pregnancy before 20 weeks' gestational age.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with history of one fresh embryo transfer failure
2. Patients with Primary infertility
3. Patients with at least one embryo with excellent quality

Exclusion Criteria:

1. Female age over 40 years old 2- Severe male factor (Azoospermia) 3- Endometriosis diagnosis and the presence of hydrosalpinges 4- Uterine factor ( polyps, myoma and previous myomectomy, …) 5- Patients with polycystic ovarian syndrome diagnosis 6- Cases with pre-implantation genetic diagnosis (PGD)indication 7- Cases with difficult embryo transfer or use of Tenaculum 8- Patients with repeated implantation failures and repeated miscarriages. 9- Female smokers

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2014-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 4 weeks
  Evaluation the rate of clinical pregnancy 4-6 weeks after embryo transfer

SECONDARY OUTCOMES:
Ongoing pregnancy | 20 weeks
  Evaluation the Ongoing pregnancy 20 weeks after pregnancy
early miscarriage rate | 12 weeks
  Evaluation thepregnancy loss under 12 weeks of gestational age
Chemical pregnancy rate | 2 weeks
  Evaluation the Chemical pregnancy rate 2 weeks after embryo transfer.
Late miscarriage rate20 weeks | 20 weeks
  Evaluation the pregnancy loss under 20 weeks of gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Maryam Hafezi, MD, Study Director — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Tahereh Madani, MD, Study Director — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Arezoo Arabipour, MSC, Principal Investigator — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Hafezi M, Madani T, Arabipoor A, Zolfaghari Z, Sadeghi M, Ramezanali F. The effect of intrauterine human chorionic gonadotropin flushing on live birth rate after vitrified-warmed embryo transfer in programmed cycles: a randomized clinical trial. Arch Gynecol Obstet. 2018 Jun;297(6):1571-1576. doi: 10.1007/s00404-018-4752-2. Epub 2018 Apr 6. PMID 29626233
- See also: Related Info — http://royaninstitute.org
- See also: Publication — https://doi.org/10.1007/s00404-018-4752-2